CLINICAL TRIAL: NCT05874830
Title: The Optimal Route of Fecal Microbiota Transplantation for Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Kimmo Salminen, MD, Specialist in Gastroenterology and Geriatrics, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T109/2021
Record Dates: First submitted 2022-04-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: IBS - Irritable Bowel Syndrome; Microbial Substitution
Keywords: IBS; FMT; Fecal microbiota transplant; microbiome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Double blinded plasebo controlled study with two treatment cohorts and one plasebo cohort
Who Masked: Participant, Care Provider, Investigator
Masking Description: The patient and the endoscopists are blinded when the FMT/plasebo is given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMT through colonoscopy (Active Comparator): Patient gets FMT in ceacum and plasebo in duodenum.
  Interventions: Other: Fecal microbiota transplant or plasebo through endoscopy
- FMT through duodenogastroscopy (Active Comparator): Patient gets plasebo in ceacum and FMT in duodenum.
  Interventions: Other: Fecal microbiota transplant or plasebo through endoscopy
- Plasebo (Placebo Comparator): Patient gets plasebo in colonoscopy and in gastroscopy.
  Interventions: Other: Fecal microbiota transplant or plasebo through endoscopy

INTERVENTIONS:
Other: Fecal microbiota transplant or plasebo through endoscopy — Colonoscopy and gastroscopy

SUMMARY:
The object of this study is to find out is there an optimal route for the fecal microbiata transplant (FMT) in patients that suffer from irritable bowel syndrome. The investigators compare outcomes in patients with repeated fecal microbiome samples and make symptomatic questionnaires (i.e. IBS-SSS, GSRS) to find out if there is difference in severity of symptoms compared to FMT given in duodenogastroscopy or in coloscopy.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional disorder affecting approximately 10% globally.[1] It is often referred to as benign, although, when severe, may cause significant reduction of quality of life and work absenteeism. The etiology of IBS is unknown although many theories have been proposed. Altered gut motility, epithelial hyperpermeability, low grade inflammation, visceral hypersensitivity, epigenetics and genetics, altered gut-brain interaction and psychological stressors have all been reported in patients with IBS.

Several studies have detected alterations in the gut microbiota composition between IBS patients and healthy controls, however a microbiota typical for IBS patients has not been conclusively defined.

Fecal microbiota transplantation has over 90% efficace in recurrent Clostridioides difficile infection (rCDI), for which it has been in clinical use for a decade. FMT is currently recommended after the second relapse of rCDI. FMT is recommended to be considered only in clinical trial settings for other indications than rCDI.

Randomized controlled studies in FMT for IBS have conflicting results. In studies with a single administration of FMT in colonoscopy a mild transient reduction of IBS symptoms has followed the intervention. In studies with fecal capsules there has not been any benefit observed. FMT via gastroscopy exerted a clear benefit with an up to 89.1% response rate. These surprisingly good results were thought to be contributable to careful donor selection, however the study included only one donor and no specific characteristics of microbiota were indentified of the suspected superdonor. Although all these three administration routes altered the microbiota of IBS patients towards that of the donor, a concurrent decrease in the symptoms was observed only when FMT was administered via colonoscopy or gastroscopy.

Manipulation of microbiota through FMT remains to be potential treatment option for IBS, however, several mechanistic questions await answering. Investigators do not yet know what is the component of stool which would carry the healing potential. There needs to be further research to define optimal donors as well as optimal patients who would be prone to benefit of FMT. The amount and number of FMT treatments may be a factor contributing to the outcome.

It is also undefined in which extend does the route of administration of FMT contribute to the outcome in IBS patients. Therefore, the investigators present a placebo-controlled trial "the optimal route" to provide further mechanistic knowledge of the optimal FMT protocol in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* 18-70 years
* known of Finnish language
* IBS, (new or old diagnosis according to Roma III or IV criteria), all subtypes
* Informed consent
* Moderate to severe IBS symptoms, IBS-SSS > 175

Exclusion Criteria:

* Pregnancy
* Antibiotic or probiotic treatment, on-going or previous month
* Abuse of drugs, alcohol or medications
* Other diagnosis besides IBS causing the GI symptoms, such as IBD, microscopic colitis or bile acid diarrhea

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the different routes of FMT, for alteration of gut microbiota towards that of the donor. | Microbiota is tested at prescreening visit, at the baseline and in 4, 12 and 52 weeks after FMT-procedure.
  The changes in the engraftment of specific bacteria between the active groups is of special interest, and the changes in the microbiota during the whole of study in the intervention group and in the plasebo group.

SECONDARY OUTCOMES:
The main clinical outcome is reduction of abdominal pain three months after FMT. | 3 months
  Gut pain: "Has your abdominal pain reduced after the intervention? "Broadening of diet: "Have you been able expand your diet after the intervention?" Global IBS symptoms: "reduction of IBS-SSS total score 50 points or more from the baseline value"
GI Symptoms: THE GASTROINTESTINAL SYMPTOM RATING SCALE (GSRS) | in 3 months and in 1 year points compared to baseline.
  Change in symptoms in GSRS questionnaire. Scale from 0 to 90, lower the score better the outcome.
Mood, General Anxiety-Disorder 7 - questionnaire | The change in the score of questionnaires between the baseline at 3 months and 12 months
  Mood changes in GAD -questionnaire. Aim is to lower the score in GAD-7 questionnaire.
Mood, Beck's Depression Inventory. | The change in the score of questionnaires between the baseline at 3 months and 12 months
  Mood changes in BDI -questionnaire. Score from 0-60. Aiming to lower the score in BDI-questionnaire.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed | through study completion, an average of 1 year
  Safety of FMT and endoscopic procedures, is there complications that need hospitalisation or other medical intervention for patients. Results given in numbers and differentiated between major and minor complications.
Broadening of diet | before intervention and after 3 months.
  D2D-questionnaire, that gives an overall index-value of how healthy subjects diet is, higher the value, healthier the diet.The D2D questionnaire gives on index-value from 0-100.

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Central hospital of Päijät-Häme, Lahti, Paijat-Hame Region
  - Turku university hospital, Turku, Southwest Finland
  - Helsinki University Hospital, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: No